CLINICAL TRIAL: NCT02602275
Title: Neuronal Correlates of Neurexan® Action in Mildly to Moderately Stressed Probands - A Randomized, Placebo-controlled, Double-blind, Cross-over Trial of Mode of Action and Response Prediction by Functional Magnetic Resonance Imaging MRI
Brief Title: Neuronal Correlates of Neurexan® Action in Mildly to Moderately Stressed Probands
Acronym: NEURIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biologische Heilmittel Heel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C1501; 2015-001802-32 (EudraCT Number)
Record Dates: First submitted 2015-10-28; First posted 2015-11-11 (Estimated); Results first posted 2025-05-08 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Acute Stress Reaction
Keywords: Stress, amygdala, functional MRI, Hariri paradigm, TSST
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute | interventions — neurexan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurexan first, then Placebo (Experimental): Participants received a single dose of three Neurexan tablets on trial Day 1. Following a washout period of 7 to 35 days, they received a single dose of three placebo tablets on trial Day 2.
  Interventions: Drug: Neurexan; Drug: Placebo
- Placebo first, then Neurexan (Experimental): Participants received a single dose of three Placebo tablets on trial Day 1. Following a washout period of 7 to 35 days, they received a single dose of three Neurexan tablets on trial Day 2.
  Interventions: Drug: Neurexan; Drug: Placebo

INTERVENTIONS:
Drug: Neurexan — 0.6 mg / tablet
  Other Names: Nx4
Drug: Placebo — Neurexan-matched Placebo tablet

SUMMARY:
The purpose of this study is to explore the effect of Neurexan® on the brain response when participants undergo an emotional stressful condition in verum compared to placebo.

DETAILED DESCRIPTION:
A randomized placebo-controlled, double-blind, two-period crossover study with an explorative design. 40 healthy males aged 31-59 years will be included in the study. Participant allocation to either Neurexan® or Placebo at study start is randomized with a ratio of 1:1, i.e. 20 Neurexan® first to 20 Placebo first individuals. Participants receive totally three tablets of either Neurexan® or Placebo per treatment period orally.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age between ≥31 to ≤59 years
3. Fluent in German language
4. Nonsmoker
5. Able to understand the explanations and instructions given by the study physician
6. Willing to adhere to the prohibitions and restrictions specified in this protocol
7. Healthy on the basis of clinical laboratory tests, physical examination, medical history, vital signs performed at Screening Visit
8. Magnetic Resonance Imaging (MRI) compatible
9. Participants must have signed a written informed consent document prior to any study procedure indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
10. Screening Scale for Chronic Stress of the Trier Inventory for Chronic Stress (TICS-SSCS) Score ≥ 9 and ≤ 36
11. Perceived Stress Scale (PSS) > 9

Exclusion Criteria:

1. Current or past history of psychotic features or a diagnosis of any psychiatric disorder as defined in the Diagnostic and Statistical Manual of Mental Disorder 4th edition (DSM-IV) Axis I (recurrent major depression, panic disorder, social phobia, obsessive-compulsory disorder; alcohol dependency; schizophrenia and mania)
2. History of depressive episodes during the last 3 months prior to Screening Visit
3. Use of any psychotropic medication or suffering from severe psychiatric illness during the last 3 months prior to Screening Visit
4. Intake of prescription drugs for sleeping disorders or nervousness within one month prior to Screening Visit
5. Intake of over the counter (OTC) medication for the treatment of sleeping disorders or nervousness within the last (one) week prior to Screening Visit
6. High chronic stress as verified with the TICS-SSCS (> 36)
7. Low chronic stress as verified with the TICS-SSCS (< 9) and PSS ≤ 9
8. Participants with Blood Pressure (BP) ≥ 160/100 on day 0 and at randomization
9. Participants with treated hypertension
10. Known allergies and/or hypersensitivity to ingredients of Neurexan® (Passiflora incarnata, Avena sativa, Coffea arabica, Zincum isovalerianicum, lactose monohydrate, magnesium stearate) or Placebo (Lactose monohydrate, magnesium stearate)
11. Known Lactose intolerance
12. Use of any psychological stress-management intervention within the last 4 weeks prior to Screening Visit
13. History of substance, drug, including nicotine, or alcohol abuse within the preceding 3 months prior to Screening Visit
14. Alcohol, drug, nicotine intake within the last 24 hours before day 0 and at randomization - confirmed by positive screening tests
15. Body Mass Index (BMI) > 30 kg/m2
16. Works regularly nights shifts
17. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic or hematologic disease as defined by clinical screening interview
18. Any somatic disease or other condition the Investigator or their duly assigned representatives believes could affect the ability of the individual to complete the study or the interpretation of the study results
19. Participants with medical illness that may have influenced brain morphology and/or physiology (e.g. uncontrolled hypertension, diabetes)
20. Participants with a history of one or more seizures without a clear and resolved aetiology
21. Participants with claustrophobia
22. Participants with tinnitus
23. Clinically significant acute illness within 7 days prior to randomization
24. Presence of metallic (ferromagnetic) implants (heart pacemaker, aneurysm clips), tattoos or piercings
25. Have received an experimental drug or used an experimental medical device (participation in any other clinical trial) within the last 30 days before study inclusion
26. Participants whose ability to speak for themselves lacks or can be doubted

Ages: 31 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Walter, PD Dr Med., Principal Investigator — Clinical Affective Neuroimaging Laboratory, Univ. Magdeburg, Germany
Locations (1):
- Clinical Affective Neuroimaging Laboratory (CANLAB), Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Herrmann L, Vicheva P, Kasties V, Danyeli LV, Szycik GR, Denzel D, Fan Y, Meer JV, Vester JC, Eskoetter H, Schultz M, Walter M. fMRI Revealed Reduced Amygdala Activation after Nx4 in Mildly to Moderately Stressed Healthy Volunteers in a Randomized, Placebo-Controlled, Cross-Over Trial. Sci Rep. 2020 Mar 2;10(1):3802. doi: 10.1038/s41598-020-60392-w. PMID 32123197
- [Result] Chand T, Alizadeh S, Jamalabadi H, Herrmann L, Krylova M, Surova G, van der Meer J, Wagner G, Engert V, Walter M. EEG revealed improved vigilance regulation after stress exposure under Nx4 - A randomized, placebo-controlled, double-blind, cross-over trial. IBRO Neurosci Rep. 2021 Sep 25;11:175-182. doi: 10.1016/j.ibneur.2021.09.002. eCollection 2021 Dec. PMID 34729551
- [Result] Mayer K, Krylova M, Alizadeh S, Jamalabadi H, van der Meer J, Vester JC, Naschold B, Schultz M, Walter M. Nx4 Reduced Susceptibility to Distraction in an Attention Modulation Task. Front Psychiatry. 2021 Nov 29;12:746215. doi: 10.3389/fpsyt.2021.746215. eCollection 2021. PMID 34912250
- [Result] Chand T, Alizadeh S, Li M, Fan Y, Jamalabadi H, Danyeli L, Nanni-Zepeda M, Herrmann L, Van der Meer J, Vester JC, Schultz M, Naschold B, Walter M. Nx4 Modulated Resting-State Functional Connectivity Between Amygdala and Prefrontal Cortex in a Placebo-Controlled, Crossover Trial. Brain Connect. 2022 Nov;12(9):812-822. doi: 10.1089/brain.2021.0189. Epub 2022 Jun 10. PMID 35438535
- [Result] Nanni-Zepeda M, Alizadeh S, Chand T, Kasties V, Fan Y, van der Meer J, Herrmann L, Vester JC, Schulz M, Naschold B, Walter M. Trait anxiety is related to Nx4's efficacy on stress-induced changes in amygdala-centered resting state functional connectivity: a placebo-controlled cross-over trial in mildly to moderately stressed healthy volunteers. BMC Neurosci. 2022 Nov 24;23(1):68. doi: 10.1186/s12868-022-00754-4. PMID 36434512
- [Result] Herrmann L, Kasties V, Boden C, Li M, Fan Y, Van der Meer J, Vester JC, Seilheimer B, Schultz M, Alizadeh S, Walter M. Nx4 attenuated stress-induced activity of the anterior cingulate cortex-A post-hoc analysis of a randomized placebo-controlled crossover trial. Hum Psychopharmacol. 2022 Sep;37(5):e2837. doi: 10.1002/hup.2837. Epub 2022 Feb 25. PMID 35213077
- [Derived] Krylova M, Alizadeh S, Izyurov I, Teckentrup V, Chang C, van der Meer J, Erb M, Kroemer N, Koenig T, Walter M, Jamalabadi H. Evidence for modulation of EEG microstate sequence by vigilance level. Neuroimage. 2021 Jan 1;224:117393. doi: 10.1016/j.neuroimage.2020.117393. Epub 2020 Sep 21. PMID 32971266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 53 screened subjects, 40 met all eligibility criteria and were randomized.
Groups:
- Neurexan First, Then Placebo: Participants received a single dose of three Neurexan tablets on experimental Day 1. Following a washout period of 7 to 35 days, they received a single dose of three placebo tablets on experimental Day 2.
- Placebo First, Then Neurexan: Participants received a single dose of three placebo tablets on experimental Day 1. Following a washout period of 7 to 35 days, they received a single dose of three Neurexan tablets on experimental Day 2.
Period: Day 1
Arm/Group | Neurexan First, Then Placebo | Placebo First, Then Neurexan
Started | 20 | 20
Received Intervention | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Washout (7-35 Days)
Arm/Group | Neurexan First, Then Placebo | Placebo First, Then Neurexan
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0
Period: Day 2
Arm/Group | Neurexan First, Then Placebo | Placebo First, Then Neurexan
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject from the placebo-first sequence was withdrawn on Day 1 before receiving the investigational medication (no dose was administered). No baseline data were collected for this subject, leaving 19 subjects in this sequence.
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurexan First, Then Placebo | Placebo First, Then Neurexan | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 43.2 (10.0) | 43.7 (9.6) | 43.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 19 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Task Data: BOLD Activation Changes Within Amygdala During Negative Faces in the Hariri Face Matching Task Between Placebo and Neurexan Treatment
Description: The neuronal drug effect was assessed by measuring changes in amygdala activity between placebo and Neurexan using fMRI 1 hour after treatment. The left amygdala was prespecified as region of interest for emotional processing and social stress. Amygdala activation in response to negative emotional faces versus neutral forms in the Hariri task was assessed. Beta values (i.e. parameter estimates) indicate the proportion of activation explained by a variable, here negatives faces or forms. Beta values serve as index of neural activity, the higher the beta value, the higher the activity. A paired t-test analysis of extracted beta values for the left amygdala was performed comparing placebo and Neurexan treatment. Amygdala hypersensitivity to negative stimuli is associated with anxiety disorders and increased stress sensitivity, while a reduction in amygdala activation may indicate a calming or modulating effect of the intervention.
Time Frame: 1 hour after taking a single dose of Neurexan or placebo
Measure: Mean (Standard Deviation); unit: Beta value
Groups:
- Neurexan: Participants received a single dose of three tablets Neurexan on one of two trial days (Day 1 or Day 2). The Neurexan "arm" describes the Neurexan condition of crossover trial. On the other day, the same participants received Placebo.
- Placebo: Participants received a single dose of three tablets Placebo on one of two trial days (Day 1 or Day 2). The Placebo "arm" describes the Placebo condition of crossover trial. On the other day, the same participants received Neurexan.
Arm/Group | Neurexan | Placebo
Number analyzed (Participants) | 39 | 39
Beta value | 0.196 (0.045) | 0.361 (0.040)
Statistical Analysis 1: Comparison: Neurexan vs Placebo; Test type: Superiority; p = 0.004, Paired t-test — Significance level is 0.05, corrected for multiple comparisons in the search volume which is anatomically defined by the Automated Anatomical Labelling Atlas (AAL) coordinates

2. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Resting-State Data: Change in Global Functional Connectivity Density of the Amygdala at Rest
Description: Resting-state fMRI scans were performed before dosing and approximately 1 hour after a single dose of Neurexan or Placebo. Highly connected functional hubs were identified by global functional connectivity density (gFCD) analysis. The number of voxels with a positive rsFC larger than the predefined threshold of r > 0.6 at a whole brain level was evaluated. gFCD was calculated for each voxel as the total number of significant correlations between this voxel and all voxels in gray matter. The gFCD value in each voxel was divided by the global mean value to improve normality. The larger the number of significant correlations, the greater the gFCD strength. Changes in gFCD strength of the amygdala from pre-dose to 1-hour post-dose were compared between the Neurexan and Placebo conditions using a within-subject repeated-measures ANOVA with main effects of time (pre- vs. post-dose) and drug (placebo vs. Nx4) and their interaction (time x drug).
Time Frame: 1 hour after taking a single dose of Neurexan or placebo
Population: Of the 39 participants, 3 were excluded due to excessive micromovement artifacts, and 1 was excluded due to data corruption.
Measure: Mean (Standard Deviation); unit: normalized FCD strength
Arm/Group | Neurexan | Placebo
Number analyzed (Participants) | 35 | 35
normalized FCD strength | 0.0139 (0.1338) | -0.0073 (0.0855)
Statistical Analysis 1: Comparison: Neurexan vs Placebo; Test type: Superiority; p > 0.05, Paired t-test — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Resting-State Data: Change in Whole-Brain Functional Connectivity of the Amygdala at Rest
Description: Resting-state fMRI scans were performed before dosing and approximately 1 hour after a single dose of Neurexan or Placebo. Left centromedial amygdala (CeMA) was defined as the seed based on probabilistic cytoarchitectonic maps. The time course of the average BOLD signal within the seed was correlated with the signals in each voxel in the whole brain. The Pearson correlation coefficients were transformed to Z values (Fisher's Z), resulting in a map representing voxel-wise strength of rsFC to the seed region. Changes in left CeMA rsFC from pre-dose to post-dose, evaluated as binary connectivity coefficients, were compared between the Neurexan and Placebo conditions.
Time Frame: 1 hour after taking a single dose of Neurexan or placebo
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Binary connectivity coefficient
Arm/Group | Neurexan | Placebo
Number analyzed (Participants) | 35 | 35
Binary connectivity coefficient | -0.0127 (0.0328) | 0.0239 (0.0346)
Statistical Analysis 1: Comparison: Neurexan vs Placebo; Test type: Superiority; p < 0.001, Paired t-test — Significance level was 0.05; The outcome was deemed exploratory, as multiplicity was controlled using a priori ordered hypotheses, but the preceding endpoint was not met

4. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Resting-State Data: Baseline Activity of the Amygdala at Rest as Measured by Amplitude of Low-Frequency Fluctuations (ALFF)
Description: The time series in each voxel of the rs-fMRI data were converted to the frequency domain using a Fast Fourier Transform (FFT), and the power spectrum was obtained. The square root of the power spectrum was computed and then averaged across each predefined frequency band. This averaged square root was taken as amplitude of low frequency fluctuation (ALFF). A ratio of the power spectrum of low-frequency range to that of the entire frequency range, i.e. the fractional ALFF (fALFF), was computed. High fALFF in the amygdala may reflect hyperactivity and could serve as a marker for heightened stress sensitivity. To examine the effect of drug on rs-metrics (RS1) while taking baseline rs-metrics before drug administration (RS0) as control variable, mean fALFF values of the amygdala were compared between placebo and Neurexan.
Time Frame: 1 hour after taking a single dose of Neurexan or placebo
Measure: Mean (Standard Deviation); unit: fractional ALFF
Arm/Group | Neurexan | Placebo
Number analyzed (Participants) | 21 | 21
fractional ALFF | -0.0120 (0.02534) | 0.0007 (0.03590)
Statistical Analysis 1: Comparison: Neurexan vs Placebo; Test type: Superiority; p > 0.05, Paired t-test — [p-value comment as in outcome 1, analysis 1]

5. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Task Data: Stress Network Activation in Response to Psychosocial Stress Induction.
Description: The neuronal drug effect was assessed by measuring activity changes within a predefined stress network, comprising the anterior cingulate cortex, medial orbitofrontal cortex, hippocampus, amygdala, and hypothalamus, between placebo and Neurexan using fMRI. Stress network activation in response to psychosocial stress induced by the ScanSTRESS paradigm was assessed. Beta values (i.e. parameter estimates) indicate the proportion of activation that is explained by a variable, in this case mental rotation or simple matching of figures. Beta-estimates serve as an index of neural activity, the higher the beta value, the higher the activity. The paradigm contrast (stress-control) for each participant was taken to a second level analysis of all voxels comprised by an ACC mask. A voxelwise paired t-test, controlled for multiple comparison, compared placebo and verum conditions. The endpoint was assessed approximately 1.5 hours post-dose after a single dose of Neurexan or placebo.
Time Frame: 1.5 hours after taking a single dose of Neurexan or placebo
Population: Of the 39 participants, 3 were excluded due to excessive micromovement artifacts.
Measure: Mean (Standard Deviation); unit: Beta Estimate
Arm/Group | Neurexan | Placebo
Number analyzed (Participants) | 36 | 36
Beta Estimate | 0.02 (0.14) | 0.41 (0.14)
Statistical Analysis 1: Comparison: Neurexan vs Placebo; Test type: Superiority; p < 0.05, Paired t-test — Significance level is 0.05, corrected for multiple comparisons in the search volume which is anatomically defined by the AAL (Automated Anatomical Labelling Atlas) coordinates; The outcome was deemed exploratory, as multiplicity was controlled using a priori ordered hypotheses, but a preceding endpoint was not met

ADVERSE EVENTS:
Time Frame: 1 day for each intervention
Description: Continuous recording of all adverse events on treatment days after randomization and receipt of at least one dose of the intervention.
Groups:
- Neurexan: Participants received a single dose of three Neurexan tablets (0.6 mg / tablet) on either Day 1 or Day 2 of the trial. The Neurexan "arm" refers to the Neurexan condition in the crossover trial. On the other trial day, the same participants received Placebo.
- Placebo: Participants received a single dose of three Placebo tablets on either Day 1 or Day 2 of the trial. The Placebo "arm" refers to the Placebo condition in the crossover trial. On the other trial day, the same participants received Neurexan.
Arm/Group | Neurexan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

LIMITATIONS AND CAVEATS:
Limited to male participants with mild to moderate chronic stress.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes